CLINICAL TRIAL: NCT04129892
Title: In Favor of My Resilient Self- Effects of an Academic Course on the Emotional Resilience of Students, While Comparing Sciences and Social Studies Faculties.
Brief Title: In Favor of My Resilient Self- Effects of an Academic Course on the Emotional Resilience of Students.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tel Hai College (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Tel Hai
Record Dates: First submitted 2019-10-15; First posted 2019-10-17 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: Preventive Therapy
Keywords: Resilience; Academic course; College students

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Course participants (Experimental): Students that enroll in the Resilience-based course during their Bachelor of science or Bachelor of social studies.
  Interventions: Behavioral: "In Favor of My Resilient Self" Academic course
- Control group- no intervention (No Intervention): Students in their Bachelor of science or Bachelor of social studies that did not attend the course, but agreed to fill out the study questionnaires.

INTERVENTIONS:
Behavioral: "In Favor of My Resilient Self" Academic course — Assessing the effect of an academic course on student's emotional resilience.
  Arms: Course participants

SUMMARY:
The course " In Favor of My Resilient Self" will guide participants to develop their strength sources, as well as practice self-calming and self-controlling exercises.

The main goals of the course are to:

1. Measure the effects on the emotional resilience and confidence of participants.
2. Assess differences in the course's affect on students from the faculty of sciences compared with students from the faculty of social studies.
3. Understand the mechanisms of the effects.

Results will be measured using the study questionnaire, to be filled out by the participants before, after, and three months after the completion of the course.

DETAILED DESCRIPTION:
The online Bachelor's degree course " In Favor of My Resilient Self" provides updated information regarding the term 'emotional resilience' and its mediating factors. Through weekly lessons and assignments, it will guide participants to developing an internal perspective on their strength sources, as well as practice self-calming and self-controlling exercises.

The main goals of the course are to:

1. Measure the effects on the emotional resilience and confidence of participants.
2. Assess differences in the course's affect on students from the faculty of sciences compared with students from the faculty of social studies.
3. Understand the mechanisms of the effects.

Results will be measured using the study questionnaire, to be filled out by the participants before, after, and three months after the completion of the course. The questionnaire will include validated questionnaires with good psychometric qualities. The study protocol was approved by Tel Hai College institutional review board. All participants, in the intervention (course participants) and in the control group (students of both faculties that didn't attend the course), received information about the program and the study and were asked to provide informed consent.

ELIGIBILITY:
Inclusion Criteria:

* Students at Tel Hai College that are interested in participating in the study, and provided informed consent.

Exclusion Criteria:

* Students that did not provide informed consent to participate in the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 322 (Estimated)
Dates: Start 2019-08-03 (Actual); Primary Completion 2021-10-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in The Connor-Davidson Resilience Scale (CD-RISC) | Measured three times over six months: at baseline, after the course ends, and three months after the completion of the course, measuring a change in scores
  The CD-RISC is based on Connor and Davidson's operational definition of resilience, which is the ability to "thrive in the face of adversity." The scale includes 25 items, from 5 sub-scales:
  1. Personal competence, high standards, and tenacity
  2. Trust in one's instincts, tolerance of negative affect, and strengthening effects of stress
  3. Positive acceptance of change and secure relationships
  4. Control
  5. Spiritual influences Scoring: Scoring of the scale is based on summing the total of all items, each of which is scored from 0-4. For the CD-RISC-25, the full range is therefore from 0 to 100, with higher scores reflecting greater resilience. (Connor KM, Davidson JRT. Depression and Anxiety 2003; 18: 71-82).

SECONDARY OUTCOMES:
Change from Baseline in Sociocultural Attitudes Towards Appearance Questionnaire-4 (SATAQ-4R) | Measured three times over six months: at baseline, after the course ends, and three months after the completion of the course, measuring a change in scores
  The Sociocultural Attitudes Toward Appearance Questionnaire-4 (SATAQ-4) is a measure of internalization of appearance ideals (i.e., personal acceptance of societal ideals) and appearance pressures (i.e., pressures to achieve the societal ideal). We included 22 items from the subscales: (1) Internalization: Thin/Low Body Fat, (2) Internalization: Muscular, (3) Internalization: General Attractiveness, (4) Pressures: Media, (5) Pressures: Peers, and (6) Pressures: Significant Others. (Schaefer et al, 2017)
Change from Baseline in Rosenberg Self-Esteem Scale (RSE) | Measured three times over six months: at baseline, after the course ends, and three months after the completion of the course, measuring a change in scores
  Rosenberg Self Esteem Scale (Rosenberg, 1965)- 10 items. Scoring involves a method of combined ratings. Low self-esteem responses are "disagree" or "strongly disagree" on items 1, 3, 4, 7, 10, and "strongly agree" or "agree" on items 2, 5, 6, 8, 9.
Change from Baseline in Depression, Anxiety and Stress Scale (DASS-21) | Measured three times over six months: at baseline, after the course ends, and three months after the completion of the course, measuring a change in scores
  Depression, Anxiety and Stress Scale - 21 Items (DASS-21) The Depression, Anxiety and Stress Scale - 21 Items (DASS-21) is a set of three self-report scales designed to measure the emotional states of depression, anxiety and stress. Each of the three DASS-21 scales contains 7 items, divided into subscales with similar content. The depression scale assesses dysphoria, hopelessness, devaluation of life, self-deprecation, lack of interest / involvement, anhedonia and inertia. The anxiety scale assesses autonomic arousal, skeletal muscle effects, situational anxiety, and subjective experience of anxious affect. The stress scale is sensitive to levels of chronic nonspecific arousal. It assesses difficulty relaxing, nervous arousal, and being easily upset / agitated, irritable / over-reactive and impatient. Scores for depression, anxiety and stress are calculated by summing the scores for the relevant items.
Change from Baseline in Body Esteem Scale (BES) | Measured three times over six months: at baseline, after the course ends, and three months after the completion of the course, measuring a change in scores
  Body Esteem Scale- This questionnaire examines self-esteem of body and physical appearance and consists of 3 subscales: appearance (10 items), weight (8 items) and attribution 187 to others (5 items). Items are rated on a 5-point scale: (1) never, (2) rarely, (3) sometimes, (4) 188 often, and (5) always. A higher score indicates higher body-esteem (Mendelson, Mendelson, & White, 2001)
Change from Baseline in The Eating Attitudes Test (EAT-26) | Measured three times over six months: at baseline, after the course ends, and three months after the completion of the course, measuring a change in scores
  Eating Attitudes Test- 26 items The Eating Attitudes validated scale for children and adolescents (Maloney, McGuire, & Daniels, 1988)

CONTACTS AND LOCATIONS:
Overall Officials: Moria Golan, Prof., Principal Investigator — Tel Hai College
Locations (1):
- Tel Hai Academic College, Kiryat Shmona, North of Israel, Israel

IPD SHARING:
Plan to Share IPD: No